CLINICAL TRIAL: NCT03571620
Title: A Multicenter, Randomized, Phase 2, Double-blind, Vehicle-controlled, Parallel Group Comparison Study to Evaluate the Safety and Efficacy of Q301 Cream in Adolescents and Adults With Mild to Moderate Atopic Dermatitis
Brief Title: Safety and Efficacy Study of Q301 in Mild to Moderate Adolescents and Adults Atopic Dermatitis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Qurient Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Q301-AD-P2-US002
Record Dates: First submitted 2018-06-20; First posted 2018-06-27 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle
- 1.0% Q301 Cream (Experimental)
  Interventions: Drug: Q301 Cream
- 1.4% Q301 Cream (Experimental)
  Interventions: Drug: Q301 Cream

INTERVENTIONS:
Drug: Q301 Cream — 1.0% or 1.4% Q301 Cream
  Arms: 1.0% Q301 Cream; 1.4% Q301 Cream
Drug: Vehicle — Vehicle Control
  Arms: Vehicle

SUMMARY:
This is a randomized, double-blind, vehicle-controlled, parallel-group comparison study to evaluate the safety and efficacy of Q301 Cream vs. vehicle in adolescent and adult subjects with mild to moderate AD. Study drug (Q301 Cream or vehicle) will be administered topically twice a day for 8 consecutive weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patient, for a period of at least three months, has had a clinical diagnosis of AD according to the Hanifin and Rajka Criteria by a board certified/eligible dermatologist.
* Patient has an Investigator's Global Assessment (IGA) score of 2 or 3 corresponding to mild or moderate AD
* Patient is in good general health and free of any disease state or physical condition that might impair evaluation of AD or which, in the investigator's opinion, exposes the patient to an unacceptable risk by study participation.

Exclusion Criteria:

* Patient has used within four weeks prior to randomization, systemic treatment with: 1) corticosteroids, 2) cyclosporine, 3) other immunosuppressive treatment or any medication known to affect AD (e.g., JAK inhibitors, etc.).

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-04-21 (Actual)

PRIMARY OUTCOMES:
proportion of patients with an IGA score of 0 (clear) or 1 (almost clear) and at least a two grade improvement in IGA score | Week 8

CONTACTS AND LOCATIONS:
Locations (1):
- Wake Forest School of Medicine Department of Dermatology, Winston-Salem, North Carolina, United States